CLINICAL TRIAL: NCT01956526
Title: CORolla™ TAA for Heart Failure and Preserved Ejection Fraction and Diastolic Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CorAssist Cadiovascular Ltd. (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CLD CRL 0403
Record Dates: First submitted 2013-08-12; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Diastolic Heart Failure NYHA Class III-IV; Diastolic Dysfunction Secondary to Aortic Stenosis
Keywords: Heart Failure with Preserved Ejection Fraction (HFpEF); Diastolic Heart Failure (DHF); Diastolic Dysfunction (DD)
MeSH Terms: conditions — Heart Failure, Diastolic

ARMS (3):
- CORolla™ TAA Stand Alone (Experimental): Single arm study design including with patients with isolated HFpEF, in NYHA f. Cl. III-IV. These patients will receive the CORolla™ TAA device. For assessments of results, intra-patient comparisons of pre-procedure and follow-up data will be performed;
  Interventions: Device: CORolla™ TAA device
- AVR and CORolla™ TAA Add On group (Experimental): patients who require aortic valve replacement (AVR) due to aortic stenosis and have diastolic dysfunction will receive the CORolla™ TAA device.
  Interventions: Device: CORolla™ TAA device
- AVR and CORolla ADD On - Control (No Intervention): patients who require only the aortic valve replacement (AVR) due to aortic stenosis and have diastolic dysfunction.

INTERVENTIONS:
Device: CORolla™ TAA device
  Arms: AVR and CORolla™ TAA Add On group; CORolla™ TAA Stand Alone

SUMMARY:
The study purpose is to evaluate the safety and feasibility of the CORolla™ TAA in two treatment groups, "CORolla™ Stand-alone group" and " AVR & CORolla™ Add on group".

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria

  * Adult (age > 18 years)
  * Diagnosis of heart failure with preserved systolic function according with ESC 2008 Guidelines (ejection fraction ≥ 50%)
  * NYHA F. Class III or IV symptoms with history of previous heart failure hospitalization in the last year
  * Able to sign informed consent and return for follow-up visits.
  * No contraindication for anticoagualation and antiplatelet treatment.
  * Cardiac medications unchanged for greater than 4 weeks (not including diuretics)
  * Pulmonary Wedge pressure > 15 mmHg documented by right heart catheterization at enrollment.
* Echocardiographic criteria

  * Preserved regional wall motion (no wall motion abnormalities).
  * Left ventricular ejection fraction ≥ 50%
  * LV end-diastolic volume index (LVEDVI) <97 ml/m2.
  * Left Atrial Volume Index: (LAVi >29 ml/m2).
  * E/E' ratio ( mean of septal and lateral ) ≥12 (applicable only to patients with sinus rhythm)
  * No intra-cardiac thrombus.
  * Minimal endocardial height from Apex to Mitral Annulus ≥ 70mm.

Exclusion Criteria:

* Cardiovascular disease

  * Uncontrolled HTN defined as > 140/90 mmHg, or >160/90 mmHg for patients on 3-drug therapy
  * Current or anticipated need for ICD, currently implanted with a cardiac resynchronization device (CRT), left ventricular assist device (LVAD).
  * Within the past 3 months - Acute myocardial infarction (AMI), cerebral vascular accident (CVA), Transient Ischemic Attack (TIA) , Percutaneous coronary intervention (PCI or transmyocardial laser revascularization (TMR or PMR)
  * Valvular disease (unless add - on to aortic valve replacement due to aortic stenosis)
  * Hypertrophic cardiomiopathy
  * Pericardial disease
  * Cor pulmonale or other cause of isolated right heart failure.
  * Non reversible pulmonary hypertension.
  * Right ventricle failure or right ventricular myocardial infarction.
  * Infiltrative heart disease
* Non-cardiovascular disease

  * Non-cardiovascular condition limiting ability to assess the 6-minute hall walk test
  * Prior surgery, radiation, or thoracic surgery limiting the ability to place the device
  * Body mass index of greater than 40
  * Uncontrolled hyperglycemic status as addressed by HbA1c >8.5%
  * Asthma COPD (e.g. FEV1 <1.5 liter), or severe restrictive lung disease
  * Severe chronic renal failure indicated by MDRD GFR <30 mL/min/1.73 m2
  * Liver impairment addressed by bilirubin > 2 mg/dl and or pseudo- colinesterasis plasma concentration < 1500 IU and/or abnormal coagulative profile
  * Severe anemia addressed by Hb concentration <10 gr/l.
  * Solid organ or hematologic transplant.
  * Previous Trans Apical procedures/implantation
* Miscellaneous conditions

  * Unwilling to fulfill the protocol medication compliance, testing, and follow-up requirements
  * Co-morbid condition that in the physician's opinion would prohibit the subject's ability to meet the protocol requirements
  * Pregnancy at the time of enrollment. (Women of child bearing potential must have a negative serum pregnancy test within two weeks prior to enrollment, or be using hormonal contraceptives or intrauterine devices)
  * Enrolled in another investigational study
  * A history of alcohol abuse, drug addiction, or other psychosocial condition that would preclude successful participation, or clear judgment and informed consent in the opinion of the Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Cardiovasculare related SAEs | 12 month post surgery
  Investigational device safety with the intended study population with respect to 12 months follow up will be demonstrated using the following:
  Cardiovascular mortality and morbidity reports at 30 days post surgery.
  Serious adverse events: death, arrhythmia, CVA, AMI, bleeding and valve injury at 12 months post-surgery.

SECONDARY OUTCOMES:
feasibility | up to 36 month post surgery
  Change in Quality of Life (QoL): Minnesota Living with Heart Failure.
Feasibility | up to 36 month post surgery
  Change in NYHA f. class
Feasibility | up to 36 month post surgery
  Change in exercise capacity as measured by the Six-Minute Walk test
Feasibility | Up to 36 month post surgery
  Composite rate of HF death and re-hospitalization at 6 months and 1 year.
Feasibility | up to 36 month post surgery
  Impact of CORolla™ TAA therapy on markers of diastolic dysfunction assessed by conventional echocardiography imaging (e.g LAVI index etc)and novel approach including Tissue Doppler Imaging (TDI)
Feasibility | up to 36 month post surgery
  Change of Wedge pressure - for safety assessment and impact of CORolla™ TAA therapy on this marker of diastolic dysfunction
Feasibility | up to 36 month post surgery
  Changes in cardiac medical therapy including daily diuretic dose

OTHER OUTCOMES:
Procedural success | intra procedural
  Success of the implant surgical procedure will be determined according to Implantation Rating Questionnaire.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Spedali Civili - Brescia Hospital, Brescia
  - Multimedica, Milan

REFERENCES:
- [Background] Dickstein K, Cohen-Solal A, Filippatos G, McMurray JJ, Ponikowski P, Poole-Wilson PA, Stromberg A, van Veldhuisen DJ, Atar D, Hoes AW, Keren A, Mebazaa A, Nieminen M, Priori SG, Swedberg K; ESC Committee for Practice Guidelines (CPG). ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2008: the Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2008 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association of the ESC (HFA) and endorsed by the European Society of Intensive Care Medicine (ESICM). Eur Heart J. 2008 Oct;29(19):2388-442. doi: 10.1093/eurheartj/ehn309. Epub 2008 Sep 17. No abstract available. PMID 18799522
- [Background] Paulus WJ, Tschope C, Sanderson JE, Rusconi C, Flachskampf FA, Rademakers FE, Marino P, Smiseth OA, De Keulenaer G, Leite-Moreira AF, Borbely A, Edes I, Handoko ML, Heymans S, Pezzali N, Pieske B, Dickstein K, Fraser AG, Brutsaert DL. How to diagnose diastolic heart failure: a consensus statement on the diagnosis of heart failure with normal left ventricular ejection fraction by the Heart Failure and Echocardiography Associations of the European Society of Cardiology. Eur Heart J. 2007 Oct;28(20):2539-50. doi: 10.1093/eurheartj/ehm037. Epub 2007 Apr 11. PMID 17428822